CLINICAL TRIAL: NCT06633510
Title: Comparison of Fluid Administered According to Plethysmographic Variability Index Versus Ideal Fluid Management in Laparoscopic Trendelenburg Surgeries
Brief Title: Fluid Administered According to PVI Versus Fluid Management in Laparoscopic Trendelenburg Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ela Erdem Hıdiroglu, principal investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ANKARA ETLİK 1
Record Dates: First submitted 2024-09-02; First posted 2024-10-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Fluid Overload Without Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massimo group (Active Comparator): The patient is not given fluids until the Massimo PVI score is >25, a 300 cc fluid bolus is given when the PVI is above 25, and fluid loading is performed at an average rate until the PVI falls below 25. If the patient's Massimo PVI is below 25, restrictive fluid therapy is applied.
  Interventions: Device: massimo group
- standart group (Active Comparator): intraoperative fluid deficit is calculated according to the 4-2-1 rule by summing up the hourly basal fasting level, intraoperative losses depending on the degree of tissue trauma (1-2mlt/kg/h in small-sized surgeries, 2-4mlt/kg/h in medium-sized surgeries, 4-8mlt/kg/h in large-sized surgeries), blood losses, urine and losses from the nasogastric tube. Fluid is given in this way.
  Interventions: Other: standart group

INTERVENTIONS:
Device: massimo group — masimo is a device for the continuous noninvasive measurement of arterial hemoglobin functional oxygen saturation (SpO2), pulse rate (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index).
  Arms: Massimo group
Other: standart group — intraoperative fluid deficit is calculated according to the 4-2-1 rule by summing up the hourly basal fasting level, intraoperative losses depending on the degree of tissue trauma (1-2mlt/kg/h in small-sized surgeries, 2-4mlt/kg/h in medium-sized surgeries, 4-8mlt/kg/h in large-sized surgeries), blood losses, urine and losses from the nasogastric tube. Fluid is given in this way.
  Arms: standart group

SUMMARY:
Investigating the ideal fluid management in Trendelenburg positions during lower abdominal laparoscopic surgeries in gynecological oncology and surgical oncology patients

DETAILED DESCRIPTION:
Laparoscopic lower abdominal surgeries include carbon dioxide (CO2) insufflation and an advanced Trendelenburg position with the head down. Increased intra-abdominal pressure can reduce cardiac index and cause changes in total body fluid balance. However, the head down Trendelenburg position increases intracranial pressure and preload. According to traditional fluid management, intraoperative fluid deficit is calculated according to the 4-2-1 rule, by summing up hourly basal fasting level, intraoperative losses due to degree of tissue trauma (1-2mlt/kg/h in minor surgeries, 2-4mlt/kg/h in medium surgeries, 4-8mlt/kg/h in major surgeries), blood losses, urine and losses from nasogastric tube.

Preservation of intravascular volume and thus provision of hemodynamic stability are among the factors affecting postoperative morbidity and mortality. Some studies have shown that standard fluid therapy is more than necessary. Current guidelines recommend more restrictive approaches by ensuring hemodynamic stability. Masimo, which we also use routinely in our clinic, is a device designed for continuous noninvasive monitoring of arterial hemoglobin functional oxygen saturation (SpO2), pulse rate (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values. In our study, in the individualization of the recommended target-oriented restrictive fluid therapy in major surgeries, by comparing the calculated fluid amount with traditional fluid management with PVI values (PVI is evaluated between 0-100.

Normavolemia 15-25 low fluid responsiveness <15 high fluid responsiveness >25) and when the patient's massimo pvi score is >25, 300cc bolus fluid will be administered and fluid will be loaded at an average speed and the PVI value will be reduced below 25. When the patient's massimo PVI value is below 25, restrictive fluid therapy will be followed.(A crystalloid fluid infusion of 2 mL/kg was administered to the patients.)

The aim was to investigate the ideal fluid management in Trendelenburg positions in lower abdominal laparoscopic surgeries performed in gynecological oncology and surgical oncology patients.

ELIGIBILITY:
İnclusion Criteria:

* between the ages of 18-80
* patients with ASA score II III
* Laparoscopic lower abdominal surgery (patients undergoing gynecological oncology and surgical oncology surgery)

Exclusion Criteria:

* ASA score IV
* Patients with heart failure and chronic kidney disease
* Patients who did not agree to participate in the study
* Cases that started laparoscopically and converted to laparotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
PI (perfusion index) | ten minutes results before induction
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate (PR) beats per minute, pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PVI (pleth variability index) | ten minutes results before induction
  arterial hemoglobin functional oxygen saturation % (SpO2, pulse rate (PR) beats per minute, pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
SPO2 (hemoglobin functional oxygen saturation) | ten minutes results before induction
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate (PR) beats per minute, pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PR (pulse rate beats per minute) | ten minutes results before induction
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate (PR) beats per minute, pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PI (perfusion index) | ten minutes when c02 insufflation is performed into the abdomen
  arterial hemoglobin functional oxygen saturation (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PVI (pleth variability index) | ten minutes when c02 insufflation is performed into the abdomen
  arterial hemoglobin functional oxygen saturation (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
SPO2 (hemoglobin functional oxygen saturation) | ten minutes when c02 insufflation is performed into the abdomen
  arterial hemoglobin functional oxygen saturation (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PR (pulse rate beats per minute) | t2(ten minutes when c02 insufflation is performed into the abdomen
  arterial hemoglobin functional oxygen saturation (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PI (perfusion index) | two hours during the surgery in the trendelenburg position
  arterialhemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PVI (pleth variability index) | two hours during the surgery in the trendelenburg position
  arterialhemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
SPO2 (hemoglobin functional oxygen saturation) | two hours during the surgery in the trendelenburg position
  arterialhemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PR (pulse rate beats per minute) | two hours during the surgery in the trendelenburg position
  arterialhemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PI (perfusion index) | five minute send of surgery
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PVI (pleth variability index) | five minute send of surgery
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
SPO2 (hemoglobin functional oxygen saturation) | five minute send of surgery
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values
PR (pulse rate beats per minute) | five minute send of surgery
  arterial hemoglobin functional oxygen saturation % (SpO2), pulse rate BPM (PR), pleth variability index (PVi) and pleth respiratory rate (Rrp) PI (perfusion index) values

CONTACTS AND LOCATIONS:
Overall Officials: ELA ERDEM HIDIROGLU, Principal Investigator — ANKARA ETLİK CİTY HOSPİTAL
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Result] Ghoundiwal D, Delaporte A, Bidgoli J, Forget P, Fils JF, Van der Linden P. Effect of pneumoperitoneum on dynamic variables of fluid responsiveness (Delta PP and PVI) during Trendelenburg position. Saudi J Anaesth. 2020 Jul-Sep;14(3):323-328. doi: 10.4103/sja.SJA_737_19. Epub 2020 May 30. PMID 32934624
- [Result] Agerskov M, Thusholdt ANW, Holm-Sorensen H, Wiberg S, Meyhoff CS, Hojlund J, Secher NH, Foss NB. Association of the intraoperative peripheral perfusion index with postoperative morbidity and mortality in acute surgical patients: a retrospective observational multicentre cohort study. Br J Anaesth. 2021 Sep;127(3):396-404. doi: 10.1016/j.bja.2021.06.004. Epub 2021 Jul 3. PMID 34226038
- [Result] Yildiz GO, Hergunsel GO, Sertcakacilar G, Akyol D, Karakas S, Cukurova Z. Perioperative goal-directed fluid management using noninvasive hemodynamic monitoring in gynecologic oncology. Braz J Anesthesiol. 2022 May-Jun;72(3):322-330. doi: 10.1016/j.bjane.2021.12.012. Epub 2022 Feb 1. PMID 35121063